CLINICAL TRIAL: NCT05992974
Title: To Identify Urinary Biomarkers in the First Trimester Associated With Gestational Diabetes Mellitus [GDM] and Achieve Early Diagnosis of GDM Using Urinary Proteomic Analysis: An Observational Study
Brief Title: To Identify Urinary Biomarkers Associated With Gestational Diabetes Mellitus [GDM]
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Mudanjiang First People's Hospital (Unknown); Mudanjiang Maternal and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202303075GDM; K4087 (Other Grant/Funding Number: Peking Union Medical College Hospital)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-08

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; urinary proteomics; early prediction
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gestational diabetes mellitus(GDM) is one of the most common complications of pregnancy. The incidence of GDM is higher in Asian than in other regions, and GDM can increase the risk of a series of perinatal complications. The investigators has been committed to the early diagnosis of GDM, and several biomarkers in the first trimester and urinary proteomic markers that were associated with GDM have been found. Based on the previous work, the aim of this study was to verify the predictive ability of urinary proteomic markers for GDM that has been found in the previous study of the researchers. This study is a multi-center, prospective, and observational study. Urine samples will be collected twice, at 12 weeks and 24-28 weeks of gestation, respectively.

DETAILED DESCRIPTION:
The eligibility criteria are as follows:

1. singleton pregnant women over 18 years old;
2. gestational age less than 12 weeks;
3. regular follow-up until delivery;
4. able to understand and sign an informed consent.

The exclusion criteria of pregnant women are as follows:

1. with impaired glucose tolerance or diabetes mellitus before pregnancy;
2. severe chronic diseases or infectious diseases (e.g., liver disease, urinary system disease, cardiovascular disease, autoimmune disease, hematological disease, AIDS and other diseases before pregnancy);
3. medications other than vitamins used during pregnancy;
4. inability to understand and follow-up regularly;
5. other conditions judged by the investigators to be inappropriate for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age who are in early pregnancy(gestational age less than 12 weeks);
* Regular prenatal examination until delivery;
* Older than 18 years old;
* Obtained informed consent from participants and/or their family members.

Exclusion Criteria:

* Twins or multiple pregnancy;
* With impaired glucose tolerance or diabetes mellitus before pregnancy;
* With severe chronic diseases or infectious diseases (e.g., liver disease, urinary system disease, cardiovascular disease, autoimmune disease, hematological disease, AIDS and other diseases before pregnancy);
* Medications other than vitamins used during pregnancy;
* Inability to understand and follow-up regularly;
* Other conditions that were judged by the investigator to be ineligible for participation in the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Our study population was pregnant women in early pregnancy who regularly visited the following two medical center: Mudanjiang First People's Hospital, and Mudanjiang Maternal and Child Health Care Hospital. All pregnant women within 12 gestational weeks are eligible for enrollment, and whether entry or not depends on their own preference. There were no requirements for household registration, place of residence, and other identify informations of the enrolled women.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gestational diabetes | at 24-28 weeks of gestation
  Diagnosed by 75g-OGTT at 24-28 weeks of gestation. GDM was diagnosed according to the International Association of Diabetes and Pregnancy Study Groups (IADPSG) criterion in 2010: fasting blood glucose ≥5.1mmol/L, and/or 1-hour blood glucose ≥10.0mmol/L, and/or 2-hour blood glucose ≥8.5mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Tedros Adhanom Ghebreyesus, Principal Investigator — World Health Organization
Locations (2):
- China (2):
  - Mudanjiang First People's Hospital, Mudanjiang, Heilongjiang
  - Mudanjiang Maternal and Child Health Hospital, Mudanjiang, Heilongjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Zhao M, Guo Z, Song S, Liu S, Yuan T, Fu Y, Dong Y, Sun H, Liu X, Zhou D, Zhao W, Sun W. Urinary proteomic analysis during pregnancy and its potential application in early prediction of gestational diabetes mellitus and spontaneous abortion. Ann Transl Med. 2022 Jul;10(13):736. doi: 10.21037/atm-21-3497. PMID 35957715
- [Result] Song S, Duo Y, Zhang Y, Qiao X, Xu J, Zhang J, Peng Z, Chen Y, Nie X, Sun Q, Yang X, Wang A, Sun W, Fu Y, Dong Y, Lu Z, Yuan T, Zhao W. The Predictive Ability of Hepatic Steatosis Index for Gestational Diabetes Mellitus and Large for Gestational Age Infant Compared with Other Noninvasive Indices Among Chinese Pregnancies: A Preliminary Double-center Cohort Study. Diabetes Metab Syndr Obes. 2021 Dec 16;14:4791-4800. doi: 10.2147/DMSO.S335364. eCollection 2021. PMID 34938090
- [Result] Song S, Zhang Y, Qiao X, Duo Y, Xu J, Peng Z, Zhang J, Chen Y, Nie X, Sun Q, Yang X, Lu Z, Liu S, Zhao T, Yuan T, Fu Y, Dong Y, Zhao W, Sun W, Wang A. HOMA-IR as a risk factor of gestational diabetes mellitus and a novel simple surrogate index in early pregnancy. Int J Gynaecol Obstet. 2022 Jun;157(3):694-701. doi: 10.1002/ijgo.13905. Epub 2021 Sep 24. PMID 34449903
- [Result] Duo Y, Song S, Zhang Y, Qiao X, Xu J, Zhang J, Peng Z, Chen Y, Nie X, Sun Q, Yang X, Wang A, Sun W, Fu Y, Dong Y, Lu Z, Yuan T, Zhao W. Predictability of HOMA-IR for Gestational Diabetes Mellitus in Early Pregnancy Based on Different First Trimester BMI Values. J Pers Med. 2022 Dec 28;13(1):60. doi: 10.3390/jpm13010060. PMID 36675721
- [Result] Song S, Zhang Y, Qiao X, Duo Y, Xu J, Peng Z, Zhang J, Chen Y, Nie X, Sun Q, Yang X, Wang A, Lu Z, Sun W, Fu Y, Dong Y, Yuan T, Zhao W. ALT/AST as an Independent Risk Factor of Gestational Diabetes Mellitus Compared with TG/HDL-C. Int J Gen Med. 2022 Jan 5;15:115-121. doi: 10.2147/IJGM.S332946. eCollection 2022. PMID 35023950